CLINICAL TRIAL: NCT02387112
Title: Early Versus Emergency Left Ventricular Assist Device Implantation in Patients Awaiting Cardiac Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Heart Institute (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Helmholtz Zentrum München (Industry); University Medicine Greifswald (Other); University of Göttingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZHK VAD Study; VAD Study Germany (Other Grant/Funding Number: DZHK/BMBF Germany)
Record Dates: First submitted 2013-06-24; First posted 2015-03-12 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: End Stage Heart Disease
Keywords: End stage heart disease; Ventricular assist device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early VAD implantation (Experimental): The experimental intervention is early implantation of a left ventricular assist device (early VAD). Patients randomized to early VAD implantation will obtain a VAD within 28 days after randomization.
  Interventions: Device: Early VAD implantation
- Emergency VAD implantation (No Intervention): The control intervention is conservative heart failure treatment, with LVAD implantation in the case of worsening heart failure (emergency VAD). All patients randomized to the control intervention will be treated according to standard medical practice. In brief, these patients are closely monitored (scheduled regular visits to outpatient department depending on the patient's condition and at least every 6 months). If the condition worsens the patient may qualify for high urgency (HU) listing and/or for VAD implantation.

INTERVENTIONS:
Device: Early VAD implantation — Implantation of a left ventricular assist device
  Arms: Early VAD implantation

SUMMARY:
The aim of the study is to assess whether, in patients who are listed for cardiac transplantation in transplantable (T) status, early implantation of a left ventricular assist device is superior to the current therapeutic strategy of medical heart failure therapy and assist device implantation only after serious deterioration of the patient's condition.

DETAILED DESCRIPTION:
Heart transplantation is considered the gold-standard therapy for end-stage systolic heart failure but the shortage of donor hearts in Germany and other countries has led to widespread use of left ventricular assist devices (LVAD). Even on the transplant list, patients' condition often deteriorate due to worsening heart failure so that they need an LVAD as a bridge until transplantation. The high mortality (one in five patients on the waiting list dies within 1 year) reflects the severity of the disease. In comparison, technical progress has reduced the complication rate seen with assist devices and, according to recent data, mortality during LVAD support is low. Patient status prior to LVAD implantation is a strong indicator for postoperative outcome, i.e. patients in worse condition are more likely to develop complications. Thus, the comparison between the standard indication and early LVAD implantation (T-status) appears timely and clinically necessary.

The paucity of donor hearts necessitates the prospective evaluation of alternative treatment regimens. The aim of the study is to assess whether, in patients with end-stage heart failure awaiting cardiac transplantation, a strategy involving early LVAD implantation is superior to a strategy of conservative medical heart failure therapy and assist device implantation only after severe deterioration of heart failure.

The investigators expect to gain insights that will be trail-blazing for the future treatment of patients with heart failure on the transplantation waiting list, including aspects of their medical care. If the study hypotheses are confirmed, the treatment of these seriously ill patients could be, on the one hand, further optimized. On the other hand, positive economic effects are highly probable.

The results will form the basis of future guidelines for the treatment of this group of patients.

Thus the study will also make a contribution to solving the problem of the ever increasing number of patients on the waiting list as opposed to the decreasing willingness to donate organs for transplantation.

As a mean of quality control of the conducted study and to retrieve more data in this population all patients who fulfill the eligibility criteria of the study but do not consent to randomization are included in a standard treatment registry.

ELIGIBILITY:
Inclusion Criteria

* Patient (male or female) eligible for heart transplantation and accepted in T Status (transplantable) on the waiting list
* Age 18 to 65 years
* Signed informed consent
* >30% 1-year mortality with the Seattle Heart Failure Model (SHFM) or at least three of the following criteria (a) to (f):

  1. cardiac index (CI) <2.5 l/min/m²
  2. pulmonary capillary wedge pressure >15 mmHg
  3. maximal oxygen uptake (VO2max) ≤10.0 ml/kg/min or ≤12.0 ml/kg/min in patients intolerant of a ß-blocker
  4. ratio of minute ventilation (VE) to carbon dioxide (VCO2) production (VE/VCO2) slope of >35
  5. at least two hospitalizations for heart failure within the previous 12 months
  6. documented increase of brain natriuretic peptide (BNP) or NTproBNP levels despite optimal medical therapy

Exclusion Criteria

* Listing for transplantation of other organs in addition to heart
* Previous cardiac surgeries (other than pacemaker or ICD surgeries)
* Contraindications to assist device implantation (e.g. mechanical aortic valve, aortic insufficiency)
* Contraindications to anticoagulation
* Expected need for a right ventricular assist device/biventricular support expected (e.g. due to tricuspid valve insufficiency grade 3+, right ventricular ratio short/long axis ≥0.6, ratio of right to left ventricular end-diastolic diameter (RVEDD/LVEDD) >0.72, restrictive cardiomyopathy)
* Presence of catecholamine support or intra-aortic balloon counterpulsation (IABP)
* Overt infections
* Fixed pulmonary hypertension (i.e. pulmonary arterial pressure (PAP) >60 mmHg and mean transpulmonary gradient (TPG) >15 mmHg or pulmonary vascular resistance (PVR) >6 Wood units despite optimal medical treatment)
* Renal insufficiency (glomerular filtration rate (GFR) <30ml/min or need for hemodialysis or hemofiltration)
* Significant coagulopathies
* Systemic lupus erythematosus, sarcoid, or amyloidosis that has multisystem involvement and is still active
* Drug abuse and/or alcohol abuse
* Incompliance
* Elevated panel reactivity levels of >50 %
* Pregnancy or breast feeding in women
* Participation in other investigational trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Randomisation untill month 60 (60 months at the most, 48 months on average)
  The time to the composite end-point of all-cause death, high urgent cardiac transplantation, disabling stroke , HF hospitalizations (including emergency room HF visits >6 hrs).

SECONDARY OUTCOMES:
Stroke | Randomisation untill month 60 (60 months at the most, 48 months on average)
  Freedom from disabling and non-disabling strokes
Listing for high-urgency (HU) cardiac transplantation | Randomisation untill month 60 (60 months at the most, 48 months on average)
Number of patients with de novo right heart failure measured by decreasing right heart ejection fraction, increasing central venous pressure and/or secondary organ failure needing catecholamines and/or right ventricular circulatory support | Randomisation untill month 60 (60 months at the most, 48 months on average)
Number of patients with hospitalizations due to device failure | Randomisation untill month 60 (60 months at the most, 48 months on average)
Number of patients with adverse events due to device failure | Randomisation untill month 60 (60 months at the most, 48 months on average)
Number of device infections requiring antibiotics and/surgical intervention | Randomisation untill month 60 (60 months at the most, 48 months on average)
Number of patients with major bleedings (needing >4 Units of blood) following VAD implantation and major bleedings due to anticoagulation therapy | Randomisation untill month 60 (60 months at the most, 48 months on average)
  Bleeding needing hospitalisation, blood transfusion and/or surgical interventions
Cardiovascular Death | Randomisation untill month 60 (60 months at the most, 48 months on average)
Number of patients suffering from secondary organ failure | Randomisation untill month 60 (60 months at the most, 48 months on average)
  Time to event of renal and/or hepatic failure
Maximum oxygen uptake (VO2 max) | Measured every 6 months from randomisation untill month 60 (60 months at the most, 48 months on average)
Heart failure survival score | Measured every 6 months from randomisation untill month 60 (60 months at the most, 48 months on average)
Seattle heart failure score | Measured every 6 months from randomisation untill month 60 (60 months at the most, 48 months on average)
New York Heart Association class (NYHA) | Measured every 6 months from randomisation untill month 60 (60 months at the most, 48 months on average)
Number of patients requiring urgent VAD implantation | Randomisation untill month 60 (60 months at the most, 48 months on average)
Rate of recurrent hospitalizations | Randomisation untill month 60 (60 months at the most, 48 months on average)
Number of patients receiving a donor heart | Randomisation untill transplantation (60 months at the most, 48 months on average)
VAD explantation due to myocardial recovery | Randomisation untill month 60 (60 months at the most, 48 months on average)
  Time to event
Short Form-36 (SF-36) | Randomisation untill month 60 (60 months at the most, 48 months on average)
  Quality of life questionnaire (QoL)
Minnesota Living with heart failure questionnaire (MLHFQ) | Randomisation untill month 60 (60 months at the most, 48 months on average)
  Quality of life questionnaire (QoL)
Mini-mental state examination (MMSE) | Randomisation untill month 60 (60 months at the most, 48 months on average)
  Quality of life questionnaire (QoL)
Quality-adjusted life year (QALY) | Randomisation untill month 60 (60 months at the most, 48 months on average)

CONTACTS AND LOCATIONS:
Overall Officials: Volkmar Falk, MD, PhD, Principal Investigator — German Heart Institute Berlin Germany
Locations (18):
- Germany (18):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen - Klinik für Herz- und Gefäßchirurgie, Bad Krozingen
  - Kerckhoff Klinik Bad Nauheim, Bad Nauheim
  - Herz- und Diabeteszentrum NRW - Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen
  - Charité - Universitätsmedizin Berlin: Campus Benjamin Franklin, Berlin
  - German Heart Center Berlin, Berlin
  - Universitätsklinikum Erlangen - Herzchirurgische Klinik, Erlangen
  - Universitätsklinikum Frankfurt - Klinik für Thorax-, Herz- und thorakale Gefäßchirurgie, Frankurt Am Main
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Med. Hochschule Hannover, Klinik für Herz-, Thorax-, Transplantations- und Gefäßchirurgie, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Klinik für Herz- und Thoraxchirurgie, Jena
  - Universitätsklinikum Schleswig Holstein - Campus Kiel, Kiel
  - Heart Center Leipzig, Leipzig
  - Universitätsklinik für Herz- und Thoraxchirurgie, Magdeburg
  - Universitätsklinikum Gießen und Marburg Klinik für Herz- und thorakale Gefäßchirurgie, Marburg
  - Herzchirurgische Klinik und Poliklinik des Klinikums der Universität München - Campus Großhadern, München
  - Universitätskrankenhaus Münster, Münster